CLINICAL TRIAL: NCT05367674
Title: Summer Harvest Adventure: A Garden-based Obesity Prevention Program for Children Residing in Low-resource Communities
Acronym: SHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Spees, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-11075
Record Dates: First submitted 2022-05-03; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Childhood Obesity
Keywords: obesity; youth; garden; diet; produce
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: Phase 2 prospective randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Clinical assessments for both groups (intervention and control) will be conducted by trained personnel that are blinded to participants' treatment arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Summer Harvest Adventure (SHA) (Experimental): Remote nutrition counseling, weekly produce harvesting, group nutrition education
  Interventions: Behavioral: Summer Harvest Adventure
- My Summer Plate (MSP) (Active Comparator): Nutrition education packet
  Interventions: Behavioral: My Summer Plate (MSP)

INTERVENTIONS:
Behavioral: Summer Harvest Adventure — Biobehavioral intervention focusing on nutrition and lifestyle behaviors.
  Arms: Summer Harvest Adventure (SHA)
Behavioral: My Summer Plate (MSP) — My Summer Plate (MSP)
  Arms: My Summer Plate (MSP)

SUMMARY:
The objective of this study is to implement and test the efficacy of the "Summer Harvest Adventure," a comprehensive garden-based behavioral, social, and environmental intervention for children (ages 8-11 years) residing in low-resource communities.

DETAILED DESCRIPTION:
The investigators will conduct a 2-arm randomized controlled trial designed to determine the efficacy of a multifaceted obesity prevention and lifestyle intervention in low-resource children and parent/adult caregiver (PAC) called "Summer Harvest Adventure." A total of 240 children (ages 8-11 years) will be randomized to the garden-based intervention (SHA) or an enhanced control group (MSP). Summer Harvest Adventure includes: 1) remote and group coaching using a focused motivational interviewing approach; 2) weekly fruit, vegetable, and herb harvesting to increase summer food access; and 3) group education for children and their families in a social setting. Assessments for both groups will be collected at orientation held one week prior to the intervention (week 0), and immediately following the completion of the intervention (week 10) by trained personnel that are blinded to participants' treatment arm assignment.

ELIGIBILITY:
Inclusion Criteria:

* Children 8-11 years of age (as of June 1) from assenting and consenting families
* English-speaking families that agree to participate; 3) residents of SNAP-eligible communities in Franklin County, Ohio.

Exclusion Criteria:

* Inability to functionally participate in harvesting; accommodations can be implemented in the future for children with special needs
* Communication difficulties (e.g. severe developmental delay)
* Lack of transportation to weekly classes or harvesting activities
* Non-English speakers; because coaching and classroom-based education are all conducted in English, we will of necessity restrict to English-speakers only during this phase

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Produce intake | Baseline and 10 weeks
  Change in fruit and vegetable intake as assessed by dermal skin carotenoid scores using Ramon Spectroscopy (Pharmanex NuSkin Biophotonic Scanner model S3)

SECONDARY OUTCOMES:
Weight | Baseline and 10 weeks
  Change in weight will be recorded with a precision of 0.1 kilogram
Family engagement | Baseline and 10 weeks
  Change in family engagement as assessed by the Expressed Emotion Adjective Checklist
Blood Pressure | Baseline and 10 weeks
  Change in blood pressure will be measured using non-invasive brachial blood pressure assessment using oscillometric technology (automated devices) to obtain BP readings
Height | Baseline and 10 weeks
  Change in standing height will be measured to the nearest 1 mm using a standardized fixed stadiometer with a vertical backboard and moveable headboard
BMI percentile | Baseline and 10 weeks
  BMI will be calculated using weight (kg) divided by the square of height (m). BMI-for-age percentile growth charts will be used to measure the size and growth patterns of children in the study

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hill EB, Chen L, Bailey MT, Singh Khalsa A, Maltz R, Kelleher K, Spees CK, Zhu J, Loman BR. Facilitating a high-quality dietary pattern induces shared microbial responses linking diet quality, blood pressure, and microbial sterol metabolism in caregiver-child dyads. Gut Microbes. 2022 Jan-Dec;14(1):2150502. doi: 10.1080/19490976.2022.2150502. PMID 36457073